CLINICAL TRIAL: NCT07274748
Title: Effects of High Intensity Interval Training Versus Intermittent Functional Training on Cardiovascular Fitness, Physical Function and Cognition in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0271 Shamama Naqvi
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Cardiorespiratory fitnss ,Cognition , Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient will be allocated .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: High-Intensity Interval Training (HIIT) (Experimental): The HIIT group will engage in session of alternating high-intensity and low-intensity exercise.
  * Total Duration: 30-35 minutes per session
  * Frequency: 3 days per week (Monday, Wednesday and Friday)
  * Duration of program: 12 weeks
  * Intensity: Fastest safe walking speed or 85%-95% heart rate reserve
  * Exercise mode: Treadmill Session structure:
    1. Warm-up
       1. Activity: Light walking/jogging
       2. Duration: 5 min
       3. Intensity: Low intensity, 40-50% of maximum heart rate.
    2. Main workout: (Interval training)
       1. Repetitions: 6-10 intervals
       2. Structure:
  High-Intensity Phase:
  1. Activity: sprinting or fast running pace
  2. Duration: 5 min
  3. Intensity: 85-95% of maximum heart rate
  Recovery phase:
  1. Activity: walking/slow jogging
  2. Duration: 1-2 mins
  3. Intensity: 50-60% of max heart rate c. Interval pattern: 5 min high intensity, followed by 1-2 min recovery. d. Total High-Intensity Duration: 4x5=20 minutes e. Total Recovery Period: 4x2=8 minutes
  4. Cool Down:
     1. Activity:
  Interventions: Other: Group A: High-Intensity Interval Training (HIIT)
- Group B: Intermittent Functional Training (IFT) (Experimental): IFT group will engage in session of task-oriented exercises (3 different tasks per circuit) focused on improving functional ability.
  * Total Duration:
    30 minutes/session; 6-9 circuits of 3 minutes each
  * Frequency: 3 days per week (Monday, Wednesday and Friday)
  * Duration of program: 12 weeks.
  * Intensity: maintain heart rate 30-50 beats per minute above resting levels.
  * Exercise mode: task-oriented functional exercises such as
  * Rolling side to side on a mat
  * Moving from lying to sitting and sitting to standing
  * Stepping and transferring from standing to the floor and back
  Session structure:
  1. Warm-up
     1. Activity: Light walking/jogging
     2. Duration: 5 min
     3. Intensity: Low intensity 40-50% of maximum heart rate.
  2. Main workout: (IFT circuits)
     * Circuit 1 (3 minutes) Task 1: Rolling side to side on a mat (1 minute). Task 2: Moving from lying to sitting (1 minute). Task 3: Standing up from a chair (1 minute). Rest (30-60 seconds).
     * Circuit 2 (3 minutes):
  Task 1: Stepping onto a
  Interventions: Other: Group B: Intermittent Functional Training (IFT)

INTERVENTIONS:
Other: Group A: High-Intensity Interval Training (HIIT) — The intervention consists of HIIT protocol performed 3-5 days per week for a period of 12 weeks, focusing on either the fastest safe walking speed for mobility gains or maintaining 85%-95% of heart rate reserve or power output at 90%-100% VO2 peak. Each session should last 25-30 minutes, utilizing a burst-to-recovery ratio of 30 seconds of intense activity followed by 30-60 seconds to 3 minutes of recovery. Treadmills or recumbent steppers will be used, with careful monitoring of intensity to prevent potential hypotensive responses.
  Arms: Group A: High-Intensity Interval Training (HIIT)
Other: Group B: Intermittent Functional Training (IFT) — IFT exercises will be performed for 3-5 days per week sessions involve 6-9 circuits of task-oriented exercises lasting about 3 minutes each, designed to enhance functional ability. Each circuit combines more demanding tasks with less intense ones to maintain heart rates 30-50 beats per minute above resting levels, achieving moderate aerobic intensity for chronic stroke survivors. Exercises are tailored to individual needs and progressively increased in difficulty, including movements like rolling, transitioning between positions, and practicing stepping and transferring
  Arms: Group B: Intermittent Functional Training (IFT)

SUMMARY:
The aim of this study is to determine comparative effects of High intensity interval training versus Intermittent functional training on cardiovascular fitness, physical function and cognition in stroke.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at General Hospital Lahore over the duration of ten months enrolling six months post stroke survivors. The 52 patients will be recruited through non-probability convenience sampling technique and will be randomly assigned to either the HIIT or IFT group through online randomizer tool. Both groups will undergo a 12-week intervention, consisting of three sessions per week with alternate-day training. The HIIT group will perform three sessions per week 30 minutes in total with each session consisting of 5 min intervals at 85-95% of their maximum heart rate, with 3-minute active recovery periods, while IFT group will perform three sessions per week 30 minutes in total with each session consisting of 6-9 circuits of task-oriented exercises both including a 5-min warm-up and cool down period. Data will be collected through different assessment tools including NIHSS (The National Institutes of Health Stroke Scale) to assess the severity of stroke, 6-minute walk test (6MWT) for cardiovascular fitness, MoCA (Montreal Cognitive Assessment or The MoCA Test) for cognition and Berg-balance scale (BBS) and TUG (Time Up and Go Test) for mobility and physical function

ELIGIBILITY:
Inclusion Criteria:• Age 50-75 years

* Both male and female stroke patients are included.
* Unilateral stroke experienced greater than 6 months prior to enrollment
* NIHSS: National Institute of Health Stroke Scale (a score of 5 to 15 represents a moderate stroke)
* Able to walk 10 minutes over ground with assistive devices as needed without physical assistance
* Able to walk 3 minutes on the treadmill at greater than 0.3 mph with no aerobic exercise contraindications.
* Stable cardiovascular condition (American Heart Association class B)
* Not currently participating in formal rehabilitation.

Exclusion Criteria:• Significant resting ECG abnormalities

* Diagnosed cardiovascular abnormalities
* Evidence of myocardial ischemia or significant arrhythmia on stress test hospitalization for cardiac or pulmonary disease within the previous 3 months, pacemaker or implanted defibrillator
* Lower extremity (LE) claudication
* Unable to communicate with investigators or correctly answer consent comprehension questions
* Severe LE spasticity (Ashworth scale score >2)
* LE weight-bearing pain >4/10 on a visual analog scale.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale(NIHSS) | 12 weeks
  The National Institutes of Health Stroke Scale (NIHSS) is a graded neurological examination that assesses speech, language cognition, inattention, visual field abnormalities, motor and sensory impairments, and ataxia. The scale was developed for use in acute-stroke therapy trials and has since been widely used as a standard part of the assessment in clinical trials. The National Institutes of Health Stroke Scale (NIHSS) demonstrates high reliability and validity in assessing stroke severity. Inter-rater and intra-rater reliability coefficients typically exceed 0.90, indicating consistent scoring among different clinicians and repeated assessments. The scale shows strong construct validity, correlating well with other measures like the modified Rankin Scale and predicting outcomes, as higher NIHSS scores are linked to increased mortality and disability. With a Cronbach's alpha above 0.90, the NIHSS is recognized as an effective tool for guiding treatment decisions and assessing patien
MoCA (Montreal Cognitive Assessment ) | 12 week
  The Montreal Cognitive Assessment (MoCA) is a one-page, 30-point cognitive screening measurement scale that takes about 10 minutes to administer. There are 12 subtasks in the MoCA test that include memory, visuospatial orientation, executive functioning, phonemic fluency, and two-item abstract thinking task, attention, concentration, and working memory, language, orientation to time and place. A score of 26 is a cutoff score to differentiate between normal and abnormal. Inter-rater Reliability (0.96) Chronbach's alpha (0.79)
The 6-minute walk test (6MWT) for cardiorespiratory fitness | 12 week
  The 6-minute walk test (6MWT) is commonly used to measure cardiovascular fitness and overall functional capacity. The 6-Minute Walk Test (6MWT) has shown strong reliability and validity in stroke patients. Specifically, studies report intra-class correlation coefficients (ICCs) ranging from 0.85 to 0.95, indicating excellent intra- and inter-rater reliability. For validity, the 6MWT correlates well with other functional measures, such as the Barthel Index and the Fugl-Meyer Assessment, with correlation coefficients often exceeding 0.70. Additionally, it has been shown to predict outcomes such as mortality and functional independence post-stroke. These statistics underscore the test's utility in assessing exercise capacity and guiding rehabilitation efforts
The Timed Up and Go (TUG) test for physical function and mobility | 12 week
  The Timed Up and Go (TUG) test is a reliable and valid assessment tool for mobility and fall risk in post-stroke patients, with inter-rater reliability demonstrating Intraclass Correlation Coefficients (ICCs) between 0.95 and 0.98, and intra-rater reliability ranging from 0.91 to 0.95. It shows strong construct validity, correlating well with other functional mobility measures like the Berg Balance Scale, with coefficients often exceeding r = 0.80. Additionally, the TUG effectively predicts fall risk, with sensitivity around 85% and specificity around 90%. Overall, the TUG test is essential for evaluating mobility and guiding rehabilitation in stroke care

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah International University, Daska Kalan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fulk GD, Echternach JL, Nof L, O'Sullivan S. Clinometric properties of the six-minute walk test in individuals undergoing rehabilitation poststroke. Physiother Theory Pract. 2008 May-Jun;24(3):195-204. doi: 10.1080/09593980701588284. PMID 18569856
- [Result] Nindorera F, Nduwimana I, Sinzakaraye A, Havyarimana E, Bleyenheuft Y, Thonnard JL, Kossi O. Effect of mixed and collective physical activity in chronic stroke rehabilitation: A randomized cross-over trial in low-income settings. Ann Phys Rehabil Med. 2023 May;66(4):101704. doi: 10.1016/j.rehab.2022.101704. Epub 2022 Dec 2. PMID 36115574
- [Result] Maeneja R, Silva CR, Ferreira IS, Abreu AM. Aerobic physical exercise versus dual-task cognitive walking in cognitive rehabilitation of people with stroke: a randomized clinical trial. Front Psychol. 2023 Oct 13;14:1258262. doi: 10.3389/fpsyg.2023.1258262. eCollection 2023. PMID 37901076
- [Result] Montero-Almagro G, Bernal-Utrera C, Geribaldi-Doldan N, Nunez-Abades P, Castro C, Rodriguez-Blanco C. Influence of High-Intensity Interval Training on Neuroplasticity Markers in Post-Stroke Patients: Systematic Review. J Clin Med. 2024 Mar 29;13(7):1985. doi: 10.3390/jcm13071985. PMID 38610750
- [Result] Gjellesvik TI, Becker F, Tjonna AE, Indredavik B, Lundgaard E, Solbakken H, Brurok B, Torhaug T, Lydersen S, Askim T. Effects of High-Intensity Interval Training After Stroke (The HIIT Stroke Study) on Physical and Cognitive Function: A Multicenter Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Sep;102(9):1683-1691. doi: 10.1016/j.apmr.2021.05.008. Epub 2021 Jun 6. PMID 34102144